CLINICAL TRIAL: NCT02918552
Title: Nitrite Benefits to Mediate Fatigability in Older HFpEF Patients
Brief Title: Oral Nitrite for Older Heart Failure With Preserved Ejection Fraction
Acronym: ONOH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gladwin, Mark, MD (Individual)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Daniel Forman, MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19070450; 1R56AG051637-01A1 (NIH)
Record Dates: First submitted 2016-09-13; First posted 2016-09-29 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium Nitrite; Nitrites

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 20 or 40 mg sodium nitrite tid
  Interventions: Drug: sodium nitrite
- Control (Placebo Comparator): 20 or 40 mg placebo tid
  Interventions: Drug: Control

INTERVENTIONS:
Drug: sodium nitrite — Subjects to receive active study drug three times daily during treatment period and then post treatment testing period.
  Other Names: nitrite
  Arms: Treatment
Drug: Control — Subjects randomized to placebo to receive three times daily during treatment period and then post treatment testing period.
  Other Names: Placebo
  Arms: Control

SUMMARY:
This is a randomized double blinded controlled trial of 20-40 mg sodium nitrite tid in subjects with HFpEF. Primary outcomes are measures of physical function with non-invasive and invasive cardiopulmonary exercise testing, and fatigability, skeletal muscle bioenergetics, serology including inflammatory markers and platelet bioenergetics, quality of life measures.

DETAILED DESCRIPTION:
Age-related physiological changes predispose to heart failure with preserved ejection fraction (HFpEF). Thus, HFpEF prevalence is escalating as the older population expands. High mortality and morbidity, diminished quality of life, and spiraling healthcare costs are typical consequences, and no effective HFpEF therapy is known. Therefore, several small exercise training (ExT) trials for HFpEF stand out by showing that ExT result in improved aerobic exercise capacity and infer that ExT constitutes novel substantive therapy. Nonetheless, such benefit was evident only after months of moderate to high intensity ExT; regimens that are unfeasible for most patients. In fact, poor compliance with ExT is typical in most HFpEF patients. The investigators propose there are intrinsic physiological components of HFpEF pathophysiology that predispose to "fatigability". The investigators advance the concept of fatigability by quantifying it as a performance-based measure; i.e., subjective tiring during a standardized steady-state walking (perceived fatigability) and deterioration of self-selected walking speed over time (performance fatigability). The investigators assert that therapies to reduce fatigability will enhance HFpEF outcomes. Ongoing studies reveal pleiotropic benefits of oral inorganic nitrite (NO2), including enhanced performance of skeletal muscle (metabolism and bioenergetics) and vasomotor responses (systemic and pulmonary). The investigators' pilot work shows safety and biological efficacy of oral NO2 capsules. Thus, the investigators propose a randomized, controlled, double-blinded trial to study oral NO2 therapy in older (≥70 years) HFpEF patients. Aim 1 explores the utility of NO2 capsules to reduce perceived and performance fatigability (rated perceived exertion), improve aerobic capacity (peak oxygen uptake) and increase daily activity (accelerometry). Aim 2 delineates the mediating processes by which NO2 benefits are achieved. Skeletal muscle determinants are differentiated from the right and left heart vasomotor dynamics by integrating assessments using 31Phosphorus magnetic resonance spectroscopy and percutaneous needle muscle biopsies with those made using non-invasive and invasive cardiopulmonary exercise testing, near infrared spectroscopy and other techniques. The principal investigator is trained geriatrics and cardiology, and is solidly oriented to the dynamics of aging and cardiovascular disease (clinically and mechanistically) with particular expertise in functional assessment and skeletal muscle gene expression as determinants of performance. The investigative team provides formidable synergies that are well-suited to this translational investigation of systemic, cellular, and sub-cellular physiological dynamics. Our proposal is significant in multiple respects: 1) HFpEF is endemic with aging and constitutes a critical contemporary healthcare challenge today's growing population of older adults. 2) Fatigability is rooted in HFpEF pathophysiology, but it has not previously been addressed as a key part of management. 3) NO2 therapy is a novel and compelling therapeutic strategy. 4) Mechanisms underlying fatigability are clarified; we advance principles of patient-centered care by clarifying mechanisms that underlie a patient's experience of fatigability.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* Diagnosis of HFpEF [adapted from the 2016 European Society of Cardiology (ESC) Guidelines to include:

  1. Prior diagnosis of HF via one of these:
* medical record diagnosis by attending cardiologist
* verbal confirmation of HFpEF with attending cardiologist
* PI review of medical record to confirm HFpEF AND 2. Ejection Fraction % ≥40
* Clinically stable (euvolemic; baseline heart rate <100 bpm) and without hospitalization or invasive cardiac procedure for 6 weeks
* Patients using 81 milligram (mg) aspirin (ASA) will be eligible, but will be asked to hold the medication for 3 days prior to biopsy. This technique has previously been used with consistent safety. Patients will also be asked to avoid non-steroidal anti-inflammatory medications (NSAIDs) for 2 days prior to the biopsy.
* Patients using anti-thrombin and anti-platelet therapy will plan to modify prior to muscle biopsies individually in coordination with the participant's primary cardiologist.

Exclusion Criteria:

* Allergy to lidocaine
* BP >180/95 or <100/60
* Anemia: Hgb<11.0 (♂),10.0 (♀)
* Dementia or inability to give informed consent
* End-stage malignancy
* Severe orthopedic exercise limitation
* Use of chronic oral corticosteroids or other medications that affect muscle function.
* Chronic alcohol or drug dependency.
* Any bleeding disorder that would contraindicate biopsy such as history of clinically significant bleeding diathesis (e.g., Hemophilia A or B, Von Willebrand's Disease or congenital Factor VII deficiency).
* Psychiatric hospitalization within the last 3 months
* Major cardiovascular event or procedure within the prior 6 weeks
* HF secondary to significant uncorrected primary valvular disease (except mitral regurgitation secondary to left ventricular dysfunction). If valve replacement has been performed, patient may not be enrolled for 12 months after this procedure.
* Severe uncorrected primary valvular heart disease (if valve replacement has been performed, patients will not be eligible for at least 12 months)
* Mechanical valve replacement requiring warfarin
* Peripheral or pulmonary artery disease
* Currently taking clopidogrel for a recent stent placement and/or a complex atherosclerotic lesion such that holding clopidogrel creates disproportionate risk.
* Current use of organic nitrates or phosphodiesterase type 5 inhibitors (PDE5s)
* Unable to hold warfarin or use bridging therapy, or to hold aspirin for 3 days (81 mg), 3 days (325 mg) prior to muscle biopsy or thienopyridine medications for 5 days prior to muscle biopsy.
* Subjects with diabetes whose HgbA1c >10.0
* Other chronic unstable disease such as active neoplasm, end stage chronic kidney, liver or other organ disease,

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Forman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Montefiore Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other future investigators as research questions arise.
Time Frame: A limit in time frame for sharing has not been defined.
Access Criteria: Only de-identified data approved for sharing by the PI.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Nitrite: 20 or 40 mg sodium nitrite tid
  sodium nitrite: Subjects to receive active study drug three times daily during treatment period and then post treatment testing period.
- Placebo: 20 or 40 mg placebo tid
  Control: Subjects randomized to placebo to receive three times daily during treatment period and then post treatment testing period.
Period: Overall Study
Arm/Group | Sodium Nitrite | Placebo
Started | 7 | 8
Completed | 6 | 6
Not Completed | 1 | 2
Not completed — Failed Pharmacokinetics | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Nitrite | Placebo | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.1 (6.2) | 74.6 (3.5) | 75.7 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
Ejection Fraction [Mean (Standard Deviation); unit: Percentage of blood] | 50.9 (10.1) | 54.8 (9.7) | 51.4 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Cardiorespiratory Fitness
Description: Assessment of peak Oxygen uptake (VO2) maximum via symptom limited exercise testing
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Population: In the treatment arm, a subject withdrew after pre-treatment testing.
  1 subject from the control arm withdrew after randomization but before testing. A second withdrew prior after pre-treatment testing, but before post-treatment testing.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 7 | 7
ml/kg/min
  VO2 at Rest, last 30 sec, Pre-treatment | 4.1 (1.5) | 4.0 (0.5)
  VO2 at Rest, last 30 sec, Post-treatment: number analyzed (Participants) | 6 | 6
  VO2 at Rest, last 30 sec, Post-treatment | 5.1 (1.0) | 4.5 (0.8)
  VO2 at Peak Exercise, last 30 sec, Pre-treatment | 18.6 (4.3) | 19.0 (3.9)
  VO2 at Peak Exercise, last 30 sec, Post-treatment: number analyzed (Participants) | 6 | 6
  VO2 at Peak Exercise, last 30 sec, Post-treatment | 19.6 (7.9) | 15.9 (7.7)
  VO2 at Peak Exercise, last 30 sec, change: number analyzed (Participants) | 6 | 6
  VO2 at Peak Exercise, last 30 sec, change | 1.4 (5.2) | -3.4 (5.2)

2. Secondary Outcome: Perceived Fatigability
Description: Assessment of Rate of Perceived Exertion (RPE) during steady state exercise testing at the last minute of the test. The RPE scale (Rate of Perceived Exertion) goes from 6-20 with a higher number indicating more effort and possibly a worse outcome.
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 7 | 7
Units on a scale
  RPE during last minute of the test, Pre-treatment | 9.1 (2.6) | 10.8 (4.0)
  RPE during last minute of the test, Post-treatment: number analyzed (Participants) | 6 | 6
  RPE during last minute of the test, Post-treatment | 8.3 (1.5) | 10.3 (3.3)
  RPE during last minute of the test, Change: number analyzed (Participants) | 6 | 6
  RPE during last minute of the test, Change | -1.2 (2.0) | -0.2 (1.6)

3. Secondary Outcome: Bioenergetics: In-Vivo 31P MRS Respirations
Description: Phosphocreatine reuptake after exercise during the kicking exercise in the 31P MRS (magnetic resonance spectroscopy)
Time Frame: Week 3 (pre drug) to week 10(post drug); approx. 8 weeks
Population: Magnetic resonance spectroscopy equipment had unexpected limited availability, which is why so few participants were analyzed.
Measure: Mean (Standard Deviation); unit: 1/s
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 2 | 1
1/s
  K PCr, Pre-treatment | .028 (.003) | .019 (0)
  K PCr, Post-treatment | .028 (.011) | .022 (0)

4. Secondary Outcome: Bioenergetics: Ex-Vivo Mitochondrial Respiration Analysis
Description: Mitochondrial respiration was analyzed by assessing O2 consumption by skeletal muscle mitochondria at Energetic State 3.1 using the Oroboros instrument. This state is generally used a marker for mitochondrial efficiency. Increases in consumption are generally linked to a better outcome.
Time Frame: Week 5 (pre-drug) to week 16 (post-drug); approx. 8 weeks
Population: Smaller amount of subjects were analyzed due to unexpected problems with specialized testing equipment availability.
Measure: Mean (Standard Deviation); unit: pmol/(s*mg)
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 4 | 5
pmol/(s*mg)
  O2 Consumption, Pre-treatment | 34.6 (16.5) | 57.7 (14.8)
  O2 Consumption, Post-treatment | 61.6 (36.2) | 46.0 (20.0)
  O2 Consumption, Overall change | 27.1 (27.4) | -11.7 (11.3)

5. Secondary Outcome: Exercise-induced Changes in Pulmonary Arterial Pressure
Description: Pulmonary arterial pressure, an indication of cardiopulmonary hemodynamics and cardiac function, was measured at rest and at peak exercise during an invasive cardiopulmonary exercise test.
Time Frame: Week 3 (pre-drug) to week 10 (post drug); approx 8 weeks
Population: Smaller amount of subjects were analyzed due to unexpected problems with specialized testing equipment availability.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 2 | 3
mmHg
  mPAP at Rest, Pre-treatment | 11.0 (4.2) | 16.0 (2.0)
  mPAP at Rest, Post-treatment | 17.5 (7.8) | 15.3 (1.5)
  mPAP at Peak Exercise, Pre-treatment | 28.5 (5.0) | 41.7 (15.1)
  mPAP at Peak Exercise, Post-treatment | 29.0 (1.4) | 34.7 (13.7)

6. Secondary Outcome: Exercise-induced Changes in Pulmonary Capillary Wedge Pressure
Description: Pulmonary capillary wedge pressure, an indication of cardiopulmonary hemodynamics and cardiac function, was measured at rest and at peak exercise during an invasive cardiopulmonary exercise test.
Time Frame: Week 3 (pre-drug) to week 10 (post drug); approx 8 weeks
Population: Smaller amount of subjects were analyzed due to unexpected problems with specialized testing equipment availability.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 2 | 3
mmHg
  PCWP at Rest, Pre-treatment | 5.5 (0.7) | 8.3 (2.1)
  PCWP at Rest, Post-treatment | 8.5 (12.0) | 5.7 (5.0)
  PCWP at Peak Exercise, Pre-treatment | 11.0 (0) | 22.7 (5.5)
  PCWP at Peak Exercise, Post-treatment | 11.5 (7.8) | 20.3 (10.6)

7. Secondary Outcome: Patients With Pulmonary Hypertension
Description: Right Ventricular-Pulmonary Artery Coupling, assessed by right ventricular ejection fraction (RVEF) and pulmonary artery systolic pressure (PASP), decreases with worsening right heart failure. We will be measuring this by assessing RVEF and PASP during invasive cardiopulmonary exercise testing in patients that meet criteria for pulmonary hypertension.
Time Frame: Week 3 (pre-drug) to week 10 (post drug); approx 8 weeks
Population: Smaller amount of subjects were analyzed due to unexpected problems with specialized testing equipment availability.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

8. Secondary Outcome: Steps From Accelerometry Assessment of Daily Activity
Description: Actigraph device-specific activity steps on daily-wear wrist device based on movement.
Time Frame: Week 1(pre-drug) to week 16(post-drug); approx. 16 weeks
Population: Only 6 subjects in either arm had functioning accelerometers with data that could be extracted and analyzed.
Measure: Mean (Standard Deviation); unit: Counts/day
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 6 | 6
Counts/day
  Actigraph Steps, Pre-treatment | 58399 (22586) | 54122 (14213)
  Steps, Post-treatment | 48741 (25534) | 53757 (18107)
  Steps, Change | -9657 (30110) | -366 (18251)

9. Secondary Outcome: Sedentary Events From Accelerometry Assessment of Daily Activity
Description: Assessment of daily activity using accelerometry on a daily-wear wrist device.
  Sedentary bout is a triggered stint of time that the patient is not moving or has low level of activity sensed by the accelerometer.
Time Frame: Week 1(pre-drug) to week 16(post-drug); approx. 16 weeks
Population: Only 6 subjects in either arm had functioning accelerometers with data that could be extracted and analyzed.
Measure: Mean (Standard Deviation); unit: bouts/day
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 6 | 6
bouts/day
  # of sedentary bouts/day, Pre-treatment | 29.7 (28.5) | 24.0 (17.2)
  # of sedentary bouts/day, Post-treatment | 23.7 (27.6) | 24.7 (24.3)
  # of sedentary bouts/day, Change | -6.0 (31.3) | 0.7 (17.4)

10. Secondary Outcome: Light Activity Duration From Accelerometry Assessment of Daily Activity
Description: Assessment of daily activity using accelerometry on a daily-wear wrist device.
  Light activity is a triggered stint of time that the patient has a slightly elevated amount of activity based on biometrics such as movement and heart rate.
Time Frame: Week 1(pre-drug) to week 16(post-drug); approx. 16 weeks
Population: Only 6 subjects in either arm had functioning accelerometers with data that could be extracted and analyzed.
Measure: Mean (Standard Deviation); unit: seconds/day
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 6 | 6
seconds/day
  Light activity (sec/day), Pre-treatment | 3288 (715) | 3317 (340)
  Light activity (sec/day), Post-treatment | 2866 (501) | 3224 (793)
  Light activity (sec/day), Change | -422 (903) | -94 (814)

11. Secondary Outcome: Moderate to Vigorous Physical Activity From Accelerometry Assessment of Daily Activity
Description: Assessment of daily activity using accelerometry on a daily-wear wrist device.
  MVPA is Moderate-to-vigorous physical activity that is a triggered stint of time that the patient has a slightly elevated amount of activity based on biometrics such as movement and heart rate.
Time Frame: Week 1(pre-drug) to week 16(post-drug); approx. 16 weeks
Population: Only 6 subjects in either arm had functioning accelerometers with data that could be extracted and analyzed.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 6 | 6
minutes/day
  MVPA, Pre-treatment | 719.3 (597.1) | 545.8 (237.3)
  MVPA, Post-treatment | 507.8 (456.3) | 548.2 (255.3)
  MVPA, Change | -211.5 (589.9) | 2.333 (254.4)

12. Secondary Outcome: Vector Magnitude Counts From Accelerometry Assessment of Daily Activity
Description: Assessment of daily activity using accelerometry on a daily-wear wrist device.
  Vector Magnitude in counts per day are accelerations in 3 dimensions that indicate activity. More counts is associated with more activity. More counts in a shorter duration of time indicate light, moderate, and vigorous activity.
Time Frame: Week 1(pre-drug) to week 16(post-drug); approx. 16 weeks
Population: Only 6 subjects in either arm had functioning accelerometers with data that could be extracted and analyzed.
Measure: Mean (Standard Deviation); unit: Counts/day
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 6 | 6
Counts/day
  Vector Magnitude, Pre-treatment | 1192.5 (379.5) | 1205 (205)
  Vector Magnitude, Post-treatment | 1043 (357) | 1122.7 (318.5)
  Vector Magnitude, Change | -149.4 (329) | -82.3 (337.3)

13. Other Pre Specified Outcome: Adiponectin
Description: Change in adiponectin
Time Frame: Week 5 (pre drug) to week 16 (post drug); approx. 8 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Blood Nitrate
Description: Change in blood levels to assess efficacy of study drug
Time Frame: Week 5 (pre drug) to week 16 (post drug); approx. 8 week
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Brain Natriuretic Protein
Description: Change in brain natriuretic protein (BNP)
Time Frame: Week 5 (pre drug) to week 16 (post drug); approx. 8 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Cardiopulmonary Exercise Testing: iCPET
Description: Invasive cardiopulmonary exercise testing
Time Frame: Week 3 (pre-drug) to week 10 (post drug); approx. 8 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Cardiopulmonary Exercise Testing; nCPET
Description: Non-invasive cardiopulmonary exercise testing
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Cognitive Function
Description: Change in pre and post scores on the Montreal Cognitive Assessment
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Co-morbid Illness
Description: Change in pre and post scores on the Charlson Comorbidity Index
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Co-morbidity Medications
Description: Medications for comorbidity managment
Time Frame: Week 1 pre drug to week 16 post drug
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Echocardiogram
Description: Change in cardiac strain
Time Frame: Week 1 pre-drug to week 16 post drug
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Fatigability
Description: Change in pre and post scores on the Pittsburgh Fatigability Index
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Frailty Index Assessment
Description: Physician assessment of frailty using the Canadian Clinical Frailty Scale
Time Frame: Week 1 screening pre-drug to week 16 post drug
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Gene Expression
Description: Change in DNA from Polymerase Chain Reaction analysis
Time Frame: Week 5 (pre drug) to week 16 (post drug); approx. 8 week
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Glomerular Filtration Rate
Description: Change in glomerular filtration rate (GFR)
Time Frame: Week 5 (pre drug) to week 16 (post drug); approx. 8 week
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Glycosylated Hemoglobin
Description: Change in glycosylated hemoglobin (HgbA1c)
Time Frame: Week 5 (pre drug) to week 16 (post drug); approx. 8 week
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Hematocrit
Description: Change in hematocrit
Time Frame: Week 1 pre drug to week 16 post drug
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Hemoglobin
Description: Change in hemoglobin
Time Frame: Week 1 pre drug to week 16 post drug
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Hemodynamics; Blood Pressure
Description: Change in Blood pressure
Time Frame: Week 1 pre drug to week 16 post drug
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Hemodynamics; Heart Rate
Description: Change in heart rate
Time Frame: Week 1 pre drug to week 16 post drug
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Muscle Protein
Description: Change in protein content of muscle fiber
Time Frame: Week 5 (pre drug) to week 16 (post drug); approx. 8 week
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Near Infrared Spectroscopy
Description: Assessment of blood flow during exercise
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Pain
Description: Change in pre and post scores on the McGill Pain Questionnaire
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Physical Frailty and Balance
Description: Change in score on Standard Physical Performance Battery at visit 2 pre drug and visit 5
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Physical Activity
Description: Change in pre and post scores on the CHAMPS (Community Healthy Activities Program for Seniors) Activities Questionnaire for Older Adults-physical activity
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Quality of Life
Description: Change in pre and post scores on the Kansas City Cardiomyopathy Questionnaire subject self reported responses
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Submaximal Exercise Performance
Description: Change in distance on six minute walk test
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Self-efficacy
Description: Change in pre and post scores on the Sullivan Cardiac Self Efficacy questionnaire
Time Frame: Week 2(pre drug) to Week 10( post drug); approx. 8 weeks
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Thyroid Stimulating Hormone
Description: Change in thyroid stimulating hormone (TSH)
Time Frame: Week 5 (pre drug) to week 16 (post drug); approx. 8 weeks
Reporting Status: Not Posted

40. Secondary Outcome: Sedentary Event Duration From Accelerometry Assessment of Daily Activity
Description: as for outcome 9
Time Frame: Week 1(pre-drug) to week 16(post-drug); approx. 16 weeks
Population: Only 6 subjects in either arm had functioning accelerometers with data that could be extracted and analyzed.
Measure: Mean (Standard Deviation); unit: minutes/bout
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 6 | 6
minutes/bout
  Average Sedentary Bout Duration, Pre | 14.8 (3) | 13.6 (2.3)
  Average Sedentary Bout Duration, Post | 14.4 (2.2) | 12.0 (6.0)
  Average Sedentary Bout Duration, Chg | -0.4 (2.4) | -1.6 (4.9)

41. Secondary Outcome: Light Activity Events Percentage of Day From Accelerometry Assessment of Daily Activity
Description: as for outcome 10
Time Frame: Week 1(pre-drug) to week 16(post-drug); approx. 16 weeks
Population: Only 6 subjects in either arm had functioning accelerometers with data that could be extracted and analyzed.
Measure: Mean (Standard Deviation); unit: % of day
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 6 | 6
% of day
  % in Light Activity, Pre-Treatment | .320 (.041) | .359 (.026)
  % in Light Activity, Post-Treatment | .306 (.033) | .359 (.327)
  % in Light Activity,Change | -0.014 (0.046) | -0.033 (0.078)

42. Secondary Outcome: Moderate to Vigorous Physical Activity Percentage From Accelerometry Assessment of Daily Activity
Description: as for outcome 11
Time Frame: Week 1(pre-drug) to week 16(post-drug); approx. 16 weeks
Population: Only 6 subjects in either arm had functioning accelerometers with data that could be extracted and analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of day
Arm/Group | Sodium Nitrite | Placebo
Number analyzed (Participants) | 6 | 6
Percentage of day
  % in MVPA, Pre-treatment | 0.066 (0.041) | 0.059 (0.023)
  % in MVPA, Post-treatment | 0.054 (0.045) | 0.055 (0.025)
  % in MVPA, Change | -0.012 (0.032) | -0.004 (0.023)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire 16 weeks the subject was in the study via telephone assessment for interval histories from visits 1-7 and 7 days after visit 7.
Groups:
- Treatment Arm: 20 or 40 mg sodium nitrite tid
  sodium nitrite: Subjects to receive active study drug three times daily during treatment period and then post treatment testing period.
- Control Arm: 20 or 40 mg placebo tid
  Control: Subjects randomized to placebo to receive three times daily during treatment period and then post treatment testing period.
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 3/7 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment Arm (N=7) | Control Arm (N=8)
Low diastolic blood pressure (Cardiac disorders) | 1 (1) | 0 (0) — DBP 58-59 during pharmacokinetic testing, asymptomatic
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) — Took bicosadyl with relief
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1/2 (1) | 0/3 (0) — Small, at wrist for iCPET (not all subjects in either arm at risk)
Subconjunctival Hemorrhage (Eye disorders) | 0 (0) | 1 (1) — Asymptomatic, and 100% clear
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) — Beta blocker dose was adjusted prior to administration of study drug/placebo
Chest pain (Gastrointestinal disorders) | 0 (0) | 0 (0) — Cardiologist advised likely GI in origin, resolved with OTC antacid
Pain at Biopsy site (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) — Greater than usual. Brief episode. Resolved spontaneously without issue.
Swelling of cheeks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2)
Leg Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 0 (0) | 1 (1)
Backache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper respiratory infection-like symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (2)
Difficulty Urinating (Renal and urinary disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Unable to afford daily medications (Social circumstances) | 0 (0) | 1 (1)
Took investigational drug/placebo early (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Magnetic Resonance Spectroscopy, Oroboros, and invasive CPET equipment unexpectedly had limited availability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT02918552/Prot_SAP_000.pdf